CLINICAL TRIAL: NCT03094273
Title: Prospective Study of 2 mm Margins for the Biopsy of Dysplastic Nevi
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 12-03921
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Dysplastic Nevi
Keywords: Melanocytic neoplasm; Biopsy; Saucerization biopsy; Skin lesion
MeSH Terms: conditions — Dysplastic Nevus Syndrome; Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Saucerization biopsy — 2 mm saucerization biopsy of dysplastic nevi

SUMMARY:
Non-interventional study to evaluate the utility of removing Dysplastic Nevi with a defined 2 mm margin.

DETAILED DESCRIPTION:
This is a prospective, observational study to evaluate the utility of removing Dysplastic Nevi (DN) with a defined 2 mm margin. This is a non-interventional study that will observe the pathology results following a standard of care biopsy. Principal Investigator (PI) hypothesize that the majority of lesions removed with this technique will have margins free of nevus cells on examination of histopathological sections. Hence, pathologists will not suggest that an additional excision be performed to remove any residual nevus. PI also hypothesize that if biopsy sites are followed over time, the rate of nevus recurrence will be low, because investigators would have removed the majority, if not all of the lesion at the time of initial biopsy.

ELIGIBILITY:
Inclusion Criteria:

* All patents seen in the practices of the study physicians are eligible to participate in the study.
* Patients must be over 18 years of age.
* Patients who are able to provide informed consent.
* Patient must have a lesion in which the differential diagnosis includes a DN and for which the study dermatologist deems it is appropriate to perform a saucerization biopsy.

Exclusion Criteria:

* Patients who are less than 18 years of age.
* Patients who are unable to provide informed consent.
* Lesions for which a saucerization biopsy is impractical in the judgment of the study dermatologist based on certain clinical factors (e.g. patient on anticoagulation therapy, lesion size and/or anatomic location).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NYU Dermatology Faculty Practice
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2013-02-25 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Clear margins on the histopathological sections examined after a 2 mm saucerazation biopsy. | Up to 1 year
  2 mm saucerization biopsy

SECONDARY OUTCOMES:
Nevus recurrence rate | Up to 1 year
  To determine the rate of nevus recurrence within 1 year of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David Polsky, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- Laura & Isaac Perlmutter Cancer Center & NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Terushkin V, Ng E, Stein JA, Katz S, Cohen DE, Meehan S, Polsky D. A prospective study evaluating the utility of a 2-mm biopsy margin for complete removal of histologically atypical (dysplastic) nevi. J Am Acad Dermatol. 2017 Dec;77(6):1096-1099. doi: 10.1016/j.jaad.2017.07.016. Epub 2017 Oct 2. PMID 28982585